CLINICAL TRIAL: NCT06934005
Title: Safety and Performance of Short- and Long-term Baseplates for Attaching the UNEEG Episight Recorder - Part II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U009 Part II
Record Dates: First submitted 2025-03-12; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Following a cross-over design in Part I of the study, two of the four initial Baseplates, is tested for longer wear time (35 days) in this Part II of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-term Baseplate A and long-term Baseplate C, concomitant use (Other): All participants wore Short-term Baseplate A behind one are and long-term Baseplate C behind the other ear for 35 days.
  Interventions: Device: Baseplate type A; Device: Baseplate type C

INTERVENTIONS:
Device: Baseplate type A — Type A: Acrylate tested for 35 days behind one ear
Device: Baseplate type C — Type C: Hydrocolloid tested for 35 days behind the other ear

SUMMARY:
The purpose of this clinical investigation is to test the safety and performance of one short- and one long-term Baseplate constructed with different types of biocompatible adhesives.

DETAILED DESCRIPTION:
This clinical investigation intended to test different biocompatible adhesives over time as part of the UNEEG Episight Baseplate construction for UNEEG™ medical A/S.

The two Baseplates reported on in this registration, is a follow-up to an initial testing of four different types of adhesive i.e., four types of Baseplates.

This study is Part II of the protocol. Part I is registered: NCT05111847

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained, and letter of authority signed before any study related activities
* Are at least 18 years of age and have full legal capacity
* Healthy skin behind the ear

Exclusion Criteria:

* Pregnant or breastfeeding
* Known allergic responses to the adhesives
* Treatment with corticosteroids, either as a cream in the area behind the ear or systemically (tablet or injection) within the last month
* Subject is unable or does not have the necessary assistance to properly operate the device system

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss (TEWL) to measure skin-friendliness | 35 days
  To evaluate the skin barrier functionality (i.e., skin-friendliness) after repeated use of Baseplates (i.e., adhesives) on the skin behind the ear.
  High levels of TEWL equates to unhealthy skin = high loss of water that passes from inside a body through the epidermis.High levels of TEWL equates to unhealthy skin = high loss of water that passes from inside a body through the epidermis.

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, Dr., Study Chair — Bispebjerg Hospital
Locations (1):
- Dermato-Venerologisk Afdeling og Videncenter for Sårheling, Bispebjerg Hospital, København NV, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT06934005/Prot_000.pdf